CLINICAL TRIAL: NCT02237469
Title: Retrospective Dosimetric Study of Prone Radiotherapy for Breast Cancer
Brief Title: Prone Breast Radiotherapy Treatment Planning Observational Study
Acronym: HUGProne
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Vincent Vinh-Hung (Other)
Collaborators: Varian Medical Systems (Industry)
Responsible Party: Sponsor-Investigator, Vincent Vinh-Hung, MD, PhD, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Other Study IDs: HUG 13-184R
Record Dates: First submitted 2014-09-07; First posted 2014-09-11 (Estimated); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Breast Cancer Female
Keywords: Breast cancer; Breast conserving surgery.; Radiotherapy.; Treatment planning.; Prone.
MeSH Terms: conditions — Breast Neoplasms | interventions — Prone Position

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Prone and supine simulation: Women with breast cancer receiving simulation in prone and in supine position for adjuvant radiation treatment.
  Interventions: Radiation: Prone and supine simulation

INTERVENTIONS:
Radiation: Prone and supine simulation — Treatment planning in the two positions.

SUMMARY:
The study purpose is to evaluate whether or not clinical characteristics of women with breast cancer can predict which position for radiation treatment, prone or supine, will be associated with a dosimetry gain. Dosimetry gain in this study means the lowest radiation dose to non-target organs (heart, lungs, contralateral breast), while giving the prescribed dose to tumor bed and ipsilateral breast.

DETAILED DESCRIPTION:
Retrospectively identify women who received curative radiation treatment after breast conserving cancer surgery, in whom simulation in prone and in supine position was performed. Compare the treatment plans for doses to targets and to non-target organs, according to clinical parameters of body mass index, size of breast, location of tumor and side. Furthermore, evaluate whether a single CT slide is enough or not to predict a dosimetry advantage.

ELIGIBILITY:
Inclusion Criteria:

* Breast conserving surgery
* Adjuvant radiation treatment
* Simulation done prone and supine

Exclusion Criteria:

* Simulation in only one position

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients addressed for adjuvant radiation treatment after breast conserving surgery for breast cancer, in whom simulation was done prone and supine.
Sampling Method: Non-Probability Sample
Enrollment: 280 (Estimated)
Dates: Start 2010-09; Primary Completion 2013-04 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Radiation dose to heart and lungs | 4 months
  Computations of doses and verification of physics charts.

SECONDARY OUTCOMES:
Radiation dose to tumor bed and ipsilateral breast | 4 months
  Computations of doses and verification of physics charts.

OTHER OUTCOMES:
Numbers of patients with dosimetry gain in prone position | 2 years
  Evaluate the dosimetry gain in subgroups classified according to body mass index, size of breast, side and location of tumor.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Vinh-Hung, MD, PhD, Principal Investigator — University of Genova
Locations (1):
- Geneva University Hospitals, Geneva, Switzerland

REFERENCES:
- [Background] Dipasquale G, Wang X, Chatelain-Fontanella V, Vinh-Hung V, Miralbell R. Automatic segmentation of breast in prone position: Correlation of similarity indexes and breast pendulousness with dose/volume parameters. Radiother Oncol. 2016 Jul;120(1):124-7. doi: 10.1016/j.radonc.2016.04.041. Epub 2016 May 10. PMID 27178144
- [Background] Andrianarison VA, Laouiti M, Fargier-Bochaton O, Dipasquale G, Wang X, Nguyen NP, Miralbell R, Vinh-Hung V. Contouring workload in adjuvant breast cancer radiotherapy. Cancer Radiother. 2018 Dec;22(8):747-753. doi: 10.1016/j.canrad.2018.01.008. Epub 2018 Oct 12. PMID 30322819
- [Background] Heymann S, Dipasquale G, Nguyen NP, San M, Gorobets O, Leduc N, Verellen D, Storme G, Van Parijs H, De Ridder M, Vinh-Hung V. Two-Level Factorial Pre-TomoBreast Pilot Study of Tomotherapy and Conventional Radiotherapy in Breast Cancer: Post Hoc Utility of a Mean Absolute Dose Deviation Penalty Score. Technol Cancer Res Treat. 2020 Jan-Dec;19:1533033820947759. doi: 10.1177/1533033820947759. PMID 32940569
- [Background] Vinh-Hung V, Leduc N, Verellen D, Verschraegen C, Dipasquale G, Nguyen NP. The mean absolute dose deviation-A common metric for the evaluation of dose-volume histograms in radiation therapy. Med Dosim. 2020 Summer;45(2):186-189. doi: 10.1016/j.meddos.2019.10.004. Epub 2019 Nov 19. PMID 31757715
- [Result] Wang X, Fargier-Bochaton O, Dipasquale G, Laouiti M, Kountouri M, Gorobets O, Nguyen NP, Miralbell R, Vinh-Hung V. Is prone free breathing better than supine deep inspiration breath-hold for left whole-breast radiotherapy? A dosimetric analysis. Strahlenther Onkol. 2021 Apr;197(4):317-331. doi: 10.1007/s00066-020-01731-8. Epub 2021 Jan 8. PMID 33416915
- [Result] Fargier-Bochaton O, Wang X, Dipasquale G, Laouiti M, Kountouri M, Gorobets O, Nguyen NP, Miralbell R, Vinh-Hung V. Prone versus supine free-breathing for right-sided whole breast radiotherapy. Sci Rep. 2022 Jan 11;12(1):525. doi: 10.1038/s41598-021-04385-3. PMID 35017568